CLINICAL TRIAL: NCT04116008
Title: Evaluation of Postoperative Analgesic Effect of Ultrasound Guided Erector Spinae Plane Block and Subcostal Transverse Abdominis Plane Block in Laparoscopic Cholecystectomy, Randomised Controlled Study
Brief Title: Erector Spinae Plane Block and Subcostal Transverse Abdominis Plane Block in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Omer Karaca, Director, Baskent University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: KA 19/152
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Controlled randomized study
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Block (Active Comparator): Ultrasound-guided bilateral Erector spinae plane block performed at end of the surgery with 40 ml of a bupivacaine/prilocaine mixture. Perioperative and postoperative routine analgesic protocol will be performed (consist of intravenous analgesics and intravenous patient-controlled analgesia) with no additional intervention (block) Standard Pain Followup and Monitorization will be performed.
  Interventions: Other: Standard Pain Followup and Monitorization
- Subcostal Abdominis Plane Block (Active Comparator): Ultrasound-guided bilateral STAP block performed at end of the surgery with 40 ml of a bupivacaine/prilocaine mixture. Perioperative and postoperative routine analgesic protocol will be performed (consist of intravenous analgesics and intravenous patient-controlled analgesia) with no additional intervention (block) Standard Pain Followup and Monitorization will be performed.
  Interventions: Other: Standard Pain Followup and Monitorization

INTERVENTIONS:
Other: Standard Pain Followup and Monitorization — Numeric Rating Scale (NRS) pain score will be recorded from recovery room followed by 2.-4.-6.-12.-24.hours. Intravenous meperidine administration at 0.5 mg / kg rescue analgesia was determined in patients with a NSR score of 4 and over in the postoperative collection room. It is planned that the patient will continue to follow the hourly NRS score in ward. Intramuscular diclofenac will be administered in this period if NRS 4 and if it is over, intravenous 0.5 mg / kg meperidine will be administered if NRS score is 4 or more after 2 hours. Salvage analgesic needs and times will be noted in detail, and the use of rescue analgesics, as well as NRS scores at designated hours, will be kept in a statistical evaluation.

SUMMARY:
Erector Spinae Plane Block is a newly defined regional anesthesia technique. Its use for many indications has been identified by case reports in the literature. As the investigators have considered that erector spinae plane block could be efficacious for providing postoperative analgesia in laparoscopic cholecystectomy, the investigators have implemented the application of this blockade into practice at the clinic Subcostal transverse abdominis plane block (STAP) is another regional anesthesia technic used for postoperative analgesia in laparoscopic cholecystectomy. Main purpose of this study is to compare the analgesic effect of ultrasound-guided erector spinae block and STAP in laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II-III
* Undergoing elective laparoscopic cholecystectomy

Exclusion Criteria:

* obesity
* ASA IV
* infection of the skin at the site of needle puncture area
* patients with known allergies to any of the study drugs
* coagulopathy
* recent use of analgesic drugs
* Inability to provide informed consent
* Severe kidney or liver disease
* Inability to operate PCA system
* Patient with psychiatric disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-11-10 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-12-24 (Actual)

PRIMARY OUTCOMES:
Pain Score | 24 hours
  Changes in Numeric Rating Scale (NRS) at rest and on movement will be recorded at intervals. NRS is a unidimensional measure of pain intensity in adults. The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").

SECONDARY OUTCOMES:
analgesic consumption | at PACU (postanesthetic care unit), 2nd, 4th, 6th, 12th and 24th hours
  Tramadol consumption in Patient Controlled Analgesia device and additional and rescue analgesic using
block related complication | in this block performing time, till patients anesthetized right after block procedure, at PACU, 2nd, 4th, 6th, 12th and 24th hours
  local anesthetic systemic toxicity during and after block procedure , pneumothorax and vascular puncture during block procedure
opioid complication | at PACU (postanesthetic care unit), 2nd, 4th, 6th, 12th and 24th hours
  sedation, itching, nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Halime Ozdemir, MD, Principal Investigator — Baskent University
Locations (1):
- Baskent University,Konya, Konya, Selcuklu, Turkey (Türkiye)

REFERENCES:
- [Background] Basaran B, Basaran A, Kozanhan B, Kasdogan E, Eryilmaz MA, Ozmen S. Analgesia and respiratory function after laparoscopic cholecystectomy in patients receiving ultrasound-guided bilateral oblique subcostal transversus abdominis plane block: a randomized double-blind study. Med Sci Monit. 2015 May 7;21:1304-12. doi: 10.12659/MSM.893593. PMID 25948166
- [Background] Aksu C, Gurkan Y. Ultrasound-guided bilateral erector spinae plane block could provide effective postoperative analgesia in laparoscopic cholecystectomy in paediatric patients. Anaesth Crit Care Pain Med. 2019 Feb;38(1):87-88. doi: 10.1016/j.accpm.2018.03.008. Epub 2018 Apr 6. No abstract available. PMID 29630940